CLINICAL TRIAL: NCT07089771
Title: Virtual Versus Dye-based Chromoendoscopy in Inflammatory Bowel Disease Surveillance Colonoscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Uppsala University Hospital (Other); Sahlgrenska University Hospital (Other); Falu Hospital (Other); Karolinska University Hospital (Other); Örebro University, Sweden (Other); Ersta Diakoni (Other); Saint Göran Hospital (Unknown)
Responsible Party: Principal Investigator, Olga Bednarska, Principal Investigator, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-02302-01
Record Dates: First submitted 2025-07-06; First posted 2025-07-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Inflammatory Bowel Disease (IBD); Ulcerative Colitis (Disorder); Crohns Disease; Colorectal Neoplasms
Keywords: virtual chromoendoscopy; dye-based chromoendoscopy; dysplasia detection; IBD surveillance colonoscopy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model, where participants with inflammatory bowel disease undergoing surveillance colonoscopy are randomly assigned to one of two groups: high-definition virtual chromoendoscopy (HD-VCE) or high-definition dye-based chromoendoscopy (HD-DCE). Each participant receives only one of the two interventions, and outcomes are compared between these independent groups. Randomization is performed prior to the procedure. The parallel design allows direct comparison of dysplasia detection rates between the two techniques without carryover effects, making it appropriate for evaluating the non-inferiority of HD-VCE compared to the current standard HD-DCE.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Chromoendoscopy (VCE) Group (Experimental): Participants randomized to this arm will undergo surveillance colonoscopy using high-definition virtual chromoendoscopy. This technique enhances mucosal visualization through advanced imaging technology without the use of dyes. The colonoscope's built-in virtual chromoendoscopy mode will be used to detect and characterize dysplastic lesions during withdrawal.
  Interventions: Procedure: Virtual Chromoendoscopy
- Dye-Based Chromoendoscopy (DCE) Group (Active Comparator): Participants randomized to this arm will undergo surveillance colonoscopy using high-definition dye-based chromoendoscopy. Indigo carmine dye will be sprayed segmentally on the colonic mucosa via a dye spray catheter to enhance visualization of mucosal patterns and detect dysplasia. Targeted biopsies will be taken from suspicious areas identified with dye staining.
  Interventions: Procedure: Dye-Based Chromoendoscopy

INTERVENTIONS:
Procedure: Virtual Chromoendoscopy — High-Definition Virtual Chromoendoscopy (HD-VCE):
  Surveillance colonoscopy using high-definition virtual chromoendoscopy enhances mucosal visualization through advanced imaging filters integrated into the colonoscope. This dye-free technique improves detection of dysplasia by increasing contrast and highlighting subtle mucosal patterns during withdrawal. HD-VCE reduces procedure time and eliminates risks related to dye application, offering a practical alternative to dye-based methods. Its efficacy in IBD surveillance requires further validation.
  Arms: Virtual Chromoendoscopy (VCE) Group
Procedure: Dye-Based Chromoendoscopy — High-Definition Dye-Based Chromoendoscopy (HD-DCE):
  Surveillance colonoscopy using high-definition dye-based chromoendoscopy involves segmental application of indigo carmine dye via a spray catheter. The dye enhances mucosal surface patterns, aiding dysplasia detection. HD-DCE is currently considered a gold standard in IBD surveillance due to superior dysplasia detection rates.
  Arms: Dye-Based Chromoendoscopy (DCE) Group

SUMMARY:
People with inflammatory bowel disease (IBD), such as ulcerative colitis or Crohn's disease affecting the colon, have a higher risk of developing colon cancer over time. To catch early signs of cancer, regular colonoscopies are recommended. In this study, the investigators are comparing two advanced methods of examining the colon during these surveillance colonoscopies. One method uses a special dye sprayed inside the colon to highlight abnormal areas (called dye-based chromoendoscopy). The other method uses new technology built into the camera to enhance the view without needing any dye (called virtual chromoendoscopy). Both methods use modern, high-definition equipment.

The purpose of this study is to find out if the newer, dye-free method is as good as the traditional dye method at detecting pre-cancerous changes (called dysplasia) in people with IBD.

Adults with IBD who are due for a routine surveillance colonoscopy may be invited to take part. Participants will be randomly assigned to one of the two methods. No additional procedures are involved, and only the way the colon is viewed differs. The investigators will also look at how long the procedures take, how many biopsies are needed, any complications, and how patients experience the exam. Participants will be followed over time using national health records to check for long-term outcomes.

This research will help doctors better understand which method is most effective and comfortable for patients, and may guide future recommendations for cancer screening in people with IBD.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, non-inferiority clinical trial designed to compare the diagnostic performance of two high-definition endoscopic imaging techniques used during surveillance colonoscopy in patients with longstanding inflammatory bowel disease (IBD) who are at increased risk for colorectal cancer. Participants will be randomly assigned to undergo colonoscopy using either a virtual (dye-free) chromoendoscopy method or a conventional dye-based chromoendoscopy technique. The primary objective is to evaluate whether virtual chromoendoscopy is non-inferior to dye- based chromoendoscopy in detecting dysplasia, a precancerous condition in the colon. Secondary outcomes include the number and type of lesions detected, predictive accuracy of targeted biopsies, examination times, patient-reported experience, complication rates, and biopsy frequency. Eligible participants are adults with a history of extensive colonic IBD of at least eight years, or additional high-risk factors such as primary sclerosing cholangitis or family history of colorectal cancer. Patients with previous colorectal cancer, prior colectomy, known untreated dysplasia, or contraindications to dye application will be excluded. All procedures will be performed using high-definition equipment and standardized bowel preparation protocols. The study includes long-term follow-up through national health registries to evaluate cancer outcomes and subsequent procedures at one and three years post-colonoscopy. The trial will be conducted across several academic and regional centers in Sweden, with an anticipated enrollment of approximately 480 patients to account for potential attrition. This study seeks to inform future guidelines by determining whether a less resource-intensive and potentially more patient-friendly method can provide equivalent surveillance efficacy in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and one of the criteria beneath:
* Extensive ulcerative colitis or indeterminate colitis (IBD-U), or Crohn's colitis involving at least one-third of the colon, with a disease history of at least 8 years
* IBD or IBD-U with primary sclerosing cholangitis (PSC)
* IBD or IBD-U with a family history of colorectal cancer in a first-degree relative

Exclusion Criteria:

* History of colorectal cancer or prior colectomy
* Contraindications to dye use
* Colonoscopies for therapeutic purposes
* Pregnancy
* Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with at least one dysplastic lesion detected during surveillance colonoscopy | Measured at the time of the index colonoscopy procedure (baseline) and confirmed by histopathological analysis post-procedure (up to 60 days)
  The primary endpoint is the proportion of enrolled patients in each study arm (HD-VCE and HD-DCE) who have at least one histologically confirmed dysplastic lesion (including low-grade dysplasia, high-grade dysplasia, or colorectal cancer) detected during the index surveillance colonoscopy.

SECONDARY OUTCOMES:
Number of dysplastic lesions detected per 10 minutes of withdrawal time | Measured during the index colonoscopy procedure.
  The rate of dysplastic lesions detected normalized by the colonoscope withdrawal time (number of dysplasia findings per 10 minutes) during the surveillance colonoscopy.
Positive predictive value (PPV) of targeted biopsies | Measured during the index colonoscopy and confirmed by pathology.
  The proportion of biopsies taken from suspicious lesions that are confirmed histologically as dysplastic or neoplastic.
Type and characterization of detected lesions | Assessed at the time of index colonoscopy and confirmed by pathology.
  Classification and histopathological characterization of lesions detected, including cancer, adenomas with low- or high-grade dysplasia, sessile serrated lesions (with or without dysplasia), hyperplastic polyps, inflammatory or post-inflammatory polyps, and non-dysplastic lesions.
Patient experience and satisfaction | Collected within 24-48 hours after the colonoscopy procedure.
  Self-reported patient experience and satisfaction scores collected using the validated survey Patient Experience Colonoscopy Scale (PECS), evaluating comfort and acceptability of each colonoscopy method. Survey responses are rated on a 4-point Likert scale ranging from very poor agreement to very good agreement, with higher values representing better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No